CLINICAL TRIAL: NCT01304394
Title: Safety During Use of Paediatric Triple Chamber Bag Formulas, Administered IV at a Weight Dependant Dose During 5 Consecutive Days, in Paediatric Patients up to 18 Years Requiring Parenteral Nutrition.
Brief Title: Safety During Use of Paediatric Triple Chamber Bag Formulas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Baxter Healthcare (Denis Bonnot), Baxter Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ped3CB/P01/06/Mu.B; 2007-001378-97 (EudraCT Number)
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Infant Nutrition Disorders; Infant, Premature, Diseases; Digestive System Disorders
Keywords: Parenteral Nutrition; Multi Chamber Bag
MeSH Terms: conditions — Infant Nutrition Disorders; Infant, Premature, Diseases; Digestive System Diseases; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- parenteral nutrition solution (Other)
  Interventions: Drug: Ped3CB

INTERVENTIONS:
Drug: Ped3CB — The Ped3CB is a ready to use, triple-chamber bag containing a sterile, nonpyrogenic combination of amino acids (Primene®, Baxter) with electrolytes, glucose, and lipids (ClinOleic®, Baxter) in separate compartments for intravenous (IV) PN. The dosage, frequency and duration is dependent on patient's weight, age, clinical status as well as addition energy or protein given enterally/orally.

SUMMARY:
The primary objective of this study was to provide daily information on the performance safety of the Ped3CB in practical therapeutic use in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized preterm newborn infants, term infants and toddlers, and children and adolescents requiring parenteral nutrition (PN) for at least 5 consecutive days.
* Preterm infants were to require PN representing, at baseline, 80% of total estimated nutritional needs, and patients in the other groups (term infants toddlers; children) were to require PN representing, at baseline, at least 50% of total estimated nutritional needs.
* Patient whose parents or legally authorized representative had provided signed written informed consent

Exclusion Criteria:

* Patients with a life expectancy < 6 days or with a severe illness with foreseeable intercurrent events that could jeopardize the patient's participation in the study were not included in the study.
* Patients with a diagnosis of shock, cardiac or renal failure with fluid overload, metabolic acidosis, respiratory failure, signs of sepsis, severe dyslipidemia, uncorrected metabolic disorders, severe sepsis, severe liver disease including cholestasis icterus, blood coagulation disorders and/or thrombophlebitis, acute myocardial infarction, or hypersensitivity to the active substance or any of the excipients of the test product, were not included in the study.
* Patients with specific nutritional requirements that could not be met by Ped3CB formulas were also excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 161 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Practical handling,ease of use and safety information (number of participants with adverse events) | measurements were taken on day 0-5 and up to day 10 on preterms and through 2 days after the last infusion of study product
  Practical handling and ease of use were measured with questionnaires and a VAS assessment of the Ped3CB, which was to be compared with the standard practice of the pharmacy or nursing ward at each site.
  All AEs were recorded during study treatment through 2 days after the last infusion. Vital signs and adverse events were recorded daily for the 5 days of the study in all patients and during the optional treatment period (an additional 5 days) in preterm newborn infants.

SECONDARY OUTCOMES:
nutritional intakes received, change from baseline body weight | measurements were taken on day 0-5 and up to day 10 on preterms
  Nutritional intakes, particularly the Ped3CB dose, were recorded daily during the treatment period.
  Body weight was measured and recorded daily. Changes from baseline to end of treatment were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Rigo, MD, PhD, Principal Investigator — CHR Citadelle
Locations (13):
- Belgium (2):
  - CHR Citadelle, Liège
  - CHU Tivoli La Louvière, Louvière
- France (11):
  - Hôpital HFME - Groupement Hospitalier Est, Bron
  - CHU de Nancy- Hôpital d'Enfants, Nancy
  - Maternité Régionale Adolphe Pinard, Nancy
  - CHU de Nantes, Nantes
  - Groupe Hospitalier Cochin-St Vincent de Paul, Paris
  - Hôpital Necker, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital pédiatrique Gatien de Clocheville, Tours

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765